CLINICAL TRIAL: NCT01186250
Title: Clinical Trial of Pioglitazone for Prevention of Cardiac Allograft Vasculopathy After Heart Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kiran Khush, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-05282010-6202; CTRU protocol 1314; IRB protocol 19373
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: cardiac allograft vasculopathy; pioglitazone; insulin resistance; heart transplant
MeSH Terms: conditions — Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): Pioglitazone
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 15mg pioglitazone taken daily for one month, 30mg pioglitazone taken daily for another month, 45mg pioglitazone taken daily for remaining ten months
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — placebo taken daily for one year
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the benefit of using the FDA-approved insulin-sensitizing agent, Pioglitazone, on human heart transplant recipients. The objectives of this project are to (1) determine if pioglitazone effectively treats insulin resistance in heart transplant recipients, and (2) to determine whether pioglitazone therapy after heart transplantation impacts the development or progression of cardiac allograft vasculopathy (CAV), a form of chronic rejection after heart transplantation.

DETAILED DESCRIPTION:
CAV, a rapidly progressive obliterative disease involving the graft coronary arteries, is the leading cause of morbidity and mortality beyond the first year after heart transplantation. This common complication occurs in almost half of recipients within 3 years after heart transplantation, and is associated with high rates of graft failure and mortality. Clinical care of heart transplant recipients in the current era is greatly limited by the lack of effective treatment options to prevent or retard the progression of CAV. CAV appears to be strongly associated with the state of insulin resistance, which is present in over half of heart transplant recipients and is characterized by metabolic abnormalities including glucose intolerance, dyslipidemia, endothelial dysfunction, and high levels of circulating inflammatory markers. Insulin resistance can be effectively treated with pioglitazone, a TZD compound which directly affects tissue insulin sensitivity. In this study, we will enroll 32 insulin-resistant heart transplant recipients and will randomize them to pioglitazone or placebo for a one-year period. We will determine the efficacy of pioglitazone for the treatment of insulin resistance and prevention of the development and progression of CAV after heart transplantation. The data generated from this study will provide important preliminary data for future, larger-scale clinical investigations.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant recipients, years 1-4 post-transplant
2. Age >= 18 years
3. Fasting TG/HDL ratio>=3.0 or Fasting TG>=150 mg/dL

Exclusion Criteria:

1. Diabetes mellitus
2. Severe liver dysfunction (ALT>=2.5 x upper limit of normal)
3. Severe renal dysfunction (GFR<30 or Stage IV CKD)
4. Moderate-severe fluid retention
5. Clinical or echocardiographic signs of left ventricular dysfunction
6. Contraindication to coronary angiography and/or IVUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Khush, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Double-blind randomized clinical trial of pioglitazone versus placebo from 2010 to 2013 in heart transplant recipients who were 1-4 years post-transplant.Eighteen heart transplant patients aged 22 to 72 years were randomized (9 to pioglitazone, 9 to placebo)
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 50.8 [23 to 72] | 49.2 [22 to 72] | 50.0 [22 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Insulin Levels Area Under Curve(AUC)
Description: Change from baseline in Insulin Levels During Oral Glucose Tolerance test at 1 year.
Time Frame: Baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: h*pmol/L
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 9 | 9
h*pmol/L | -47.7 [-171.3 to 75.9] | 10.7 [-76.8 to 98.2]

2. Secondary Outcome: Change in Intimal Volume
Description: Intimal volume is defined as external elastic membrane volume minus lumen (luminal) volume measured at the heart Catheterization and intravascular Ultrasound( IVUS)
Time Frame: baseline and 1 year
Population: The number of participants enrolled were not all included in the intimal volume analysis because the Angiographic diagnostic evaluation needed for intimal volume measurement was clinically inappropriate for 3 in the pioglitazone arm and 5 in the Placebo arm at 12 months post transplant.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 4
mm^3 | 12.2 (39.9) | -26.8 (46.7)

3. Secondary Outcome: Change in Levels of Fasting Glucose at Baseline and 1 Year
Description: Oral Glucose Tolerance Test : blood was drawn for fasting plasma glucose and insulin levels, followed by ingestion of a solution containing 75grams of glucose. Repeat blood samples were collected for glucose and insulin levels at 30, 90, and 120 minutes after glucose ingestion. All glucose measurements were performed by the Clinical Translational Research Unit (CTRU) Stanford University.
Time Frame: Baseline and 1 year
Population: One participant in each group did not complete the OGTT.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 8 | 8
mg/dL | 2.1 (19) | 11 (33)

4. Secondary Outcome: Change From Baseline in TG/HDL Ratio at One Year
Description: Triglyceride ratio to High Density Lipoprotien
Time Frame: Baseline and 1 year
Population: One drop out
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 8 | 8
ratio | -0.03 (6) | -1.2 (3.3)

5. Secondary Outcome: Change in Maximal Intimal Thickness(MIT) by Intravascular Unltrasound(IVUS)
Description: The change in maximal intimal thickness (MIT) from baseline to one year was recorded for several matched sites in the same coronary artery, the cross sections, predominantly in the left anterior descending coronary artery, from baseline to one-year follow-up, were studied. The IVUS cross sections were matched by using identifiable landmarks in the images, such as bifurcations or arterial calcification, or external landmarks, such as coronary veins or pericardium. In addition, the one-year IVUS studies were obtained with an angiographic roadmap of where the initial IVUS study was performed along the length of the vessel. The IVUS system auto pullback was performed at .5 mm/s from the mid-distal portion of the study vessel, where an easily identifiable landmark was visible (i.e., branchpoint). The following items were measured for each patient: maximal intimal thickness (MIT), intimal area (IA), and vessel area.
Time Frame: Baseline and 1 year
Population: number participants analyzed contained drops out due to clinical reasons
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 4
mm | -0.01 (0.3) | -0.02 (0.1)

6. Secondary Outcome: Change From Baseline in ADMA (Asymmetric Dimethylarginine) at One Year.
Description: Competitive ELISA assay in Stanford laboratory.
Time Frame: Baseline and 1 year
Population: One participant in one arm did not have Baseline or one year data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 8 | 8
umol/L | -0.05 (0.1) | -0.02 (0.1)

7. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (HsCRP) at One Year
Description: measure of low levels of C-reactive protein to identify low but persistent levels of inflammation
Time Frame: Baseline and 1 year
Population: participant drop put
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 7 | 7
mg/L | -3 (3) | 2 (4)

ADVERSE EVENTS:
Time Frame: Adverse event reporting was started at first dose and approximatly one year later ( at final dose and testing) plus 30 days.
Description: Assessment of adverse events was made by routine Comprehensive physical exam by MD, routine echocardiography, routine Comprehensive laboratory Chemistry metabolic panel, Complete Blood count, Lipid profile and all relevant drug level in the Transplant arena. In addition post GTT, research team called participant to follow up for any complaints.
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No